CLINICAL TRIAL: NCT00190983
Title: A Phase II Evaluation of Pemetrexed (Alimta) in the Treatment of Recurrent Carcinoma of the Cervix
Brief Title: A Trial for Patients With Advanced/Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Gynecologic Oncology Group (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8367; H3E-US-JMGS
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-08-24 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Cervical Intraepithelial Neoplasia; Uterine Neoplasms; Genital Neoplasms, Female
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Neoplasms; Genital Neoplasms, Female | interventions — Pemetrexed

ARMS (1):
- Pemetrexed (Experimental)
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed: 900 mg/m2 (700 mg/m2 for patients with prior radiotherapy) intravenous (IV) over 10 minutes every 21 days until disease progression.

SUMMARY:
This phase II trial is studying the antitumor activity of single agent pemetrexed 900mg/m2 IV over 10 minutes in patients with recurrent cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent squamous or non-squamous cell carcinoma of the cervix with documented disease progression
* Measurable disease
* Gynecologic Oncology Group (GOG) performance status 0-2
* Patients must have received one prior systemic chemotherapy for persistent or recurrent disease
* Patients with mild to moderate renal insufficiency should avoid taking non-steroidal anti-inflammatory drugs (NSAIDs_ with short elimination half-lives for a period of 2 days before, the day of, and 2 days following administration of pemetrexed.
* All patients taking NSAIDs with longer half-lives, should interrupt dosing for at least 5 days before, the day of, and 2 days following pemetrexed administration.
* Folic Acid (350-1000 ug) must be given daily beginning approximately 5-7 days prior to first does of pemetrexed and continuing daily until 3 weeks after the last dose of study therapy.
* Vitamin B12 (1000 ug) will be administered as an intramuscular injection approximately 1 to 2 weeks prior to first dose of pemetrexed and repeated approximately every 9 weeks until 3 weeks after the last dose of study therapy

Exclusion Criteria:

* Prior Pemetrexed
* Patients who have received radiation to more than 25% of marrow bearing areas
* Any evidence of other malignancy within last 5 years, with exception of non-melanoma skin cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Miller, MD, Study Chair — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group 215-854-0770, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pemetrexed
Started | 29
Completed | 27 (Completed means patient received treatment and was evaluable for response.)
Not Completed | 2
Not completed — Inevaluable (never treated) | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed
Number analyzed (Participants) | 27
Age, Customized [Number; unit: participants]
  <40 years | 6
  40-49 years | 9
  50-59 years | 7
  60-69 years | 4
  >69 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 24
  Black | 2
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 27
Cell Type [Number; unit: participants]
  Squamous | 19
  Adenocarcinoma | 6
  Clear cell | 1
  Adenosquamous | 1
Gynecologic Oncology Group (GOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully active | 16
    1 - Ambulatory, Restricted Strenuous Activity | 9
    2 - Ambulatory, No Work Activities | 2
Prior Therapy [Number; unit: participants]
  Prior Chemotherapy | 27
  No Prior Chemotherapy | 0
  Prior Radiotherapy | 23
  No Prior Radiotherapy | 4
Tumor Grade [Number; unit: participants] — Assesses the extent to which cancer cells are similar in appearance and function to healthy cells of the same tissue type. Grades range from 1 (least aggressive and best prognosis) to 4 (most aggressive and worst prognosis).
  participants
    G1 - Well-Differentiated | 5
    G2 - Moderately Differentiated | 15
    G3 - Poorly Differentiated | 5
    Unspecified | 2

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Best response recorded from the start of treatment until disease progression/recurrence using Response Evaluation Criteria In Solid Tumors (RECIST) criteria that defines when participants improve ("respond"), stay the same ("stable"), or worsen ("progression") during treatment.
Time Frame: baseline to measured progressive disease (up to 5 years)
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 27
participants
  Complete Response | 0
  Partial Response | 4
  Stable Disease | 16
  Disease Progression | 7

2. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause.
Time Frame: time of initial response until documented tumor progression (up to 5 years)
Population: All enrolled participants who had either a complete response (n=0) or partial response (n=4).
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 4
months | 4.4 [4.2 to 33.7]

3. Secondary Outcome: Progression-Free Survival
Description: The period from study entry until disease progression, death or date of last contact.
Time Frame: baseline until documented tumor progression (up to 5 years)
Population: All enrolled participants who experienced disease progression.
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 7
months | 3.1 [0.9 to 23.7]

4. Secondary Outcome: Overall Survival
Description: Overall survival is the duration from enrollment to death. For patients who are alive, overall survival is censored at the last contact.
Time Frame: baseline until death from any cause (up to 5 years)
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 27
months | 7.4 [1.4 to 23.7]

ADVERSE EVENTS:
Arm/Group | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 5
Other Adverse Events (participants affected / at risk) | 27
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed
Febrile neutropenia (Blood and lymphatic system disorders) | 1/27 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1/27 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/27 (1)
Pyelonephritis (Infections and infestations) | 1/27 (1)
Blood alkaline phosphatase increased (Investigations) | 1/27 (1)
Haemoglobin decreased (Investigations) | 1/27 (1)
White blood cell count decreased (Investigations) | 1/27 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1/27 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1/27 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1/27 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Pemetrexed
Anemia (Blood and lymphatic system disorders) | 23/27
Leukopenia (Blood and lymphatic system disorders) | 19/27
Lymphatics (Blood and lymphatic system disorders) | 4/27
Neutropenia (Blood and lymphatic system disorders) | 17/27
Thrombocytopenia (Blood and lymphatic system disorders) | 10/27
Cardiovascular (Cardiac disorders) | 2/27
Auditory (Ear and labyrinth disorders) | 2/27
Ocular (Eye disorders) | 4/27
Gastrointestinal (Gastrointestinal disorders) | 16/27
Nausea/vomiting (Gastrointestinal disorders) | 13/27
Constitutional (General disorders) | 21/27
Pain (General disorders) | 12/27
Hepatic (Hepatobiliary disorders) | 5/27
Infection (Infections and infestations) | 12/27
Alkaline phosphatase (Investigations) | 11/27
Serum glutamic oxaloacetic transaminase (Investigations) | 4/27
Metabolic (Metabolism and nutrition disorders) | 20/27
Neurotoxicity (Nervous system disorders) | 8/27
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 3/27
Alopecia (Skin and subcutaneous tissue disorders) | 4/27
Dermatologic (Skin and subcutaneous tissue disorders) | 11/27
Hemorrhage (Vascular disorders) | 2/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days